CLINICAL TRIAL: NCT06102902
Title: A Phase 1 Study of ZEN003694 (ZEN-3694) in Combination With Cetuximab and Encorafenib in Patients With Refractory BRAF V600E Metastatic Colorectal Cancer
Brief Title: Testing the Addition of Anti-cancer Drug, ZEN003694, to the Usual Chemotherapy Treatment, Cetuximab Plus Encorafenib, for Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-08787; NCI-2023-08787 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2024-0120; 10605 (Other: University of Texas MD Anderson Cancer Center LAO); 10605 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2023-10-25; First posted 2023-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Recurrent Colorectal Adenocarcinoma; Refractory Colorectal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; Cetuximab; (225)Ac-DOTA-c(RGDyK); encorafenib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ZEN003694, cetuximab, encorafenib) (Experimental): Patients receive ZEN003694 PO QD on days 1-28 of each cycle, cetuximab IV over 120 minutes on days 1 and 15 of each cycle, and encorafenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, CT or MRI, and collection of blood samples throughout the trial. Patients may also undergo biopsy at screening and on study.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Cetuximab; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Encorafenib; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX 818; LGX-818; LGX818
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase I trial tests the safety, best dose, and effectiveness of ZEN003694 in combination with cetuximab and encorafenib in treating patients with colorectal cancer that has not responded to previous treatment (refractory), that has come back after a period of improvement (relapsed), and that has spread from where it first started (primary site) to other places in the body (metastatic). ZEN003694 is a protein inhibitor that binds to BET proteins. When ZEN003694 binds to BET proteins, it disrupts gene expression. Preventing the expression of certain growth-promoting genes may inhibit proliferation of tumor cells that over-express BET proteins. Immunotherapy with monoclonal antibodies, such as cetuximab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Encorafenib is an enzyme inhibitor. It inhibits pathways that are responsible for controlling cell proliferation and survival, which may lead to a decrease in tumor cell proliferation. Both cetuximab and encorafenib have been approved to treat cancer. Adding ZEN003694 to cetuximab and encorafenib may be more effective at treating patients with refractory metastatic colorectal cancer than giving the usual treatment (cetuximab and encorafenib) alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of BET bromodomain inhibitor ZEN-3694 (ZEN003694) when used in combination with cetuximab and encorafenib.

II. To define the safety profile of combination of ZEN003694, encorafenib, and cetuximab.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate clinical response signals of the combination. III. To assess the pharmacodynamic (PD) profile of the combination as defined by MAPK inhibition.

EXPLORATORY OBJECTIVE:

I. To characterize pharmacodynamics and potential mechanisms of resistance to therapy via whole exome sequencing (WES), reverse phase protein array (RPPA), ribonucleic acid sequencing (RNAseq), and assay for transposase-accessible chromatin with sequencing (ATACseq)/HiSeq 4000 or NovaSeq following progression on treatment.

OUTLINE: This is a dose-escalation study of ZEN003694 followed by a dose-expansion study.

Patients receive ZEN003694 orally (PO) once daily (QD) on days 1-28 of each cycle, cetuximab intravenously (IV) over 120 minutes on days 1 and 15 of each cycle, and encorafenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multi-gated acquisition scan (MUGA), computed tomography (CT) or magnetic resonance imaging (MRI), and collection of blood samples throughout the trial. Patients may also undergo biopsy at screening and on study.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed and radiographically measurable metastatic colorectal adenocarcinoma with known BRAF V600E mutation, confirmed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory with at least one tumor measurable as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and for which standard curative or palliative measures do not exist or are no longer effective
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of ZEN003694 in combination with cetuximab and encorafenib in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin (Hb) ≥ 9 mg/dl
* Total bilirubin ≤ 1.5 mg/dl (excluding Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional upper limit of normal (ULN)
* Creatinine clearance (CrCL) glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. Patients should be New York Heart Association Functional Classification of class II or better
* Patients must have progressed after at least 1 prior systemic treatment for incurable advanced or metastatic disease
* Patients must have received prior treatment with the combination of encorafenib and cetuximab. They must have tolerated the combination at doses planned for the study
* The effects of ZEN003694 on the developing human fetus are unknown. For this reason and because BRD and BET inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 4 months following the last dose of study drug. Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of investigational product. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 or other agents used in study
* Patients with uncontrolled intercurrent illness including, but not limited to, active bleeding diatheses, poorly controlled infection/disorders, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694. As proton pump inhibitors (PPIs), H2 receptor antagonists, and antacids may alter the pharmacokinetics of ZEN003694 by reducing ZEN003694 exposure, patients receiving proton pump inhibitors are ineligible. If H2 blockers or other acid reducing agents are used concomitantly with ZEN003694, a staggered dosing schedule should be used, either dose ZEN003694 2 hours before the H2 blocker or 10-12 hours after an H2 blocker. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Pregnant women are excluded from this study because ZEN003694 is BRD and BET inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZEN003694, breastfeeding should be discontinued if the mother is treated with ZEN003694. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (dose escalation cohort) | Up to completion of dose escalation phase
  Will be determined based on the number of grade 3 or 4 adverse events in patients who participate on the study. Toxicities will be graded according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).
Recommended phase 2 dose (dose escalation cohort) | Up to completion of dose escalation phase
  Will be determined based on the number of grade 3 or 4 adverse events in patients who participate on the study. Toxicities will be graded according to CTCAE v 5.0.

SECONDARY OUTCOMES:
Time to progression | Time between consent onto study and progression, withdraw, or death, assessed up to 1 year
  Will be estimated according to Kaplan-Meier analysis.
Time to death | Time between consent onto study and death, assessed up to 1 year
  Will be estimated according to Kaplan-Meier analysis.
MAPK inhibition | Up to 1 year
  MAPK inhibition, measured by phosphorylated ERK pharmacodynamic profiling, will be evaluated to determine efficacy of the combination.

OTHER OUTCOMES:
Presence or absence of a given gene mutation | At pre-treatment and post-progression
  The presence or absence of a given gene mutation will be evaluated by next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Alonso Martinez, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (15):
- United States (15):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Lee HM, Zheng Z, Sorokin A, Wong CW, Napolitano S, Chowdhury S, Kanikarla PM, Singh AK, Kochat V, Bristow CA, Srinivasan S, Peoples M, Arslan E, Alshenaifi JY, Villarreal OE, Morris VK, Shen JP, Meric-Bernstam F, Jain AK, Fowlkes NW, Anderson A, Menter DG, Saw AK, Rai K, Kopetz S. Reprogramming of Cellular Plasticity via ETS and MYC Core-regulatory Circuits During Response to MAPK Inhibition in BRAF-mutant Colorectal Cancer. bioRxiv [Preprint]. 2025 Jun 20:2025.06.15.659716. doi: 10.1101/2025.06.15.659716. PMID 40611889